CLINICAL TRIAL: NCT01308086
Title: A Multicenter Trial Investigating the Duration of Adjuvant Therapy(3 vs. 6 Months) With the FOLFOX 4 or XELOX Regimen for Patients With High Risk Stage II or Stage III Colon Cancer
Brief Title: Adjuvant Therapy(3 vs. 6 Months) With the FOLFOX 4 or XELOX for Stage II or Stage III Colon Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hellenic Oncology Research Group (Other)
Collaborators: University Hospital of Crete (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT/09.12
Record Dates: First submitted 2011-03-01; First posted 2011-03-03 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: CRC
Keywords: Cancer; colorectal cancer; adjuvant chemotherapy; capecitabine; oxaliplatin; 5 fluorouracil
MeSH Terms: conditions — Neoplasms; Colorectal Neoplasms | interventions — Fluorouracil; Leucovorin; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FOLFOX 4 - 6months or XELOX -6months (Active Comparator)
  Interventions: Drug: 5-Fluorouracil; Drug: Leucovorin; Drug: Oxaliplatin; Drug: Capecitabine
- FOLFOX4 -3months or XELOX -3months (Experimental)
  Interventions: Drug: 5-Fluorouracil; Drug: Leucovorin; Drug: Capecitabine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: 5-Fluorouracil — 5-FU 400mg/m2 Bolus and then 22 hours 5-FU 600mg/m2 IV, days 1 & 2, q2w, for 12 cycles
  Other Names: 5-FU
  Arms: FOLFOX 4 - 6months or XELOX -6months
Drug: Leucovorin — Leucovorin 200mg/m2 IV in 2 hours, days 1 & 2, q2w, for 12 cycles
  Arms: FOLFOX 4 - 6months or XELOX -6months
Drug: Oxaliplatin — Oxaliplatin 85mg/m2 in 2 hours IV, day 1, q2w, for 12 cycles
  Other Names: LoHP
  Arms: FOLFOX 4 - 6months or XELOX -6months
Drug: Capecitabine — Capecitabine 1000 mg/m2 X 2 ,days 1-14, q2w, for 8 cycles
  Other Names: Xeloda
  Arms: FOLFOX 4 - 6months or XELOX -6months
Drug: Oxaliplatin — Oxaliplatin 130 mg/m2 in 2 hours IV, day 1, q2w, for 8 cycles
  Other Names: LoHP
  Arms: FOLFOX 4 - 6months or XELOX -6months
Drug: 5-Fluorouracil — 5-FU 400mg/m2 Bolus and then 22 hours 5-FU 600mg/m2 IV, days 1 & 2, q2w, for 6 cycles
  Other Names: 5-FU
  Arms: FOLFOX4 -3months or XELOX -3months
Drug: Leucovorin — Leucovorin 200mg/m2 IV in 2 hours, days 1 & 2, q2w, for 6 cycles
  Arms: FOLFOX4 -3months or XELOX -3months
Drug: Capecitabine — Capecitabine 1000 mg/m2 X 2 ,days 1-14, q2w, for 4 cycles
  Other Names: Xeloda
  Arms: FOLFOX4 -3months or XELOX -3months
Drug: Oxaliplatin — Oxaliplatin 130 mg/m2 in 2 hours IV, day 1, q2w, for 4 cycles
  Other Names: LoHP
  Arms: FOLFOX4 -3months or XELOX -3months
Drug: Oxaliplatin — Oxaliplatin 85mg/m2 in 2 hours IV, day 1, q2w, for 6 cycles
  Other Names: LoHP
  Arms: FOLFOX4 -3months or XELOX -3months

SUMMARY:
The purpose of this study is to compare whether a 3-month treatment is at least not inferior to a 6-month treatment (FOLFOX-4 6 vs. 12 cycles or XELOX 4 cycles vs. 8 cycles) in terms of RFS in patients with high risk stage II or stage III radically resected colon cancer.

DETAILED DESCRIPTION:
Six months of adjuvant chemotherapy with 5-FU and oxaliplatin for patients with stage III colon cancer is the world-wide standard of care, based on the MOSAIC and C-07 trials. However, it leads to significant cost, toxicity, and inconvenience. In particular, the onset of oxaliplatin induced cumulative dose-dependent neuropathies is a significant issue. The ability to maintain efficacy with a reduced duration of therapy would have clear advantage to patients, to providers, and to the health care system.

Multiple large trials in the 1990s demonstrated that the previous standard of 12 months of therapy could be reduced to 6 months. A single small trial with 5-FU alone demonstrated similar outcomes for 3 versus 6 months of therapy. Thus, it is proposed to definitively evaluate the non-inferiority of 3 months of oxaliplatin-based adjuvant chemotherapy versus the current standard of 6 months. The primary endpoint will be disease-free survival (DFS).

It is essential to have sufficient power to eliminate the possibility of clinically meaningful inferiority of 3 months of therapy: a huge number of patients will be necessary. Previous efforts and experience have conclusively demonstrated that in colon cancer, a single, global trial is impractical. Consequently, an international, prospective pooled analysis will be performed, gathering data of independent trials run in different countries, to answer the single primary hypothesis that 3 months of adjuvant therapy with FOLFOX/XELOX is non-inferior to the current standard of 6 months. Among six planned countries, the Greek intergroup will conduct one of these trials.

ELIGIBILITY:
Inclusion Criteria:

* Histologically- - confirmed adenocarcinoma of the colon or rectum stage III or stage with at least one of the follow characteristics T4 tumours, undifferentiated tumor grade >3, bowel obstruction or perforation, vascular or lymphatic or perineural invasion, <12 nodes examined, Stage IV.
* Signed written informed consent
* Randomization between 2 -8 weeks after curative surgery
* Age >18 years
* ECOG performance Status 0-1
* Pretreatment CEA within UNL
* Post-menopausal women or women willing to accept the use of an effective contraception. Pre-menopausal women should have a negative pregnancy test within 72 hours prior to randomization
* Men should also accept to use an effective contraception
* R0 resections

Exclusion Criteria:

* Evidence of metastatic disease (including presence of tumor cells in ascites or peritoneal carcinomatosis resected "en bloc")
* Evidence of other malignancies within the last 5 years (other than curatively treated basal cell carcinoma of the skin and/or in situ carcinoma of the cervix)
* No pregnant or lactating women
* Presence of clinically relevant cardiovascular disease
* Presenc of medical history or current evidence of CNS disease
* Presence of peripheral neuropathy ≤ grade 1 (CTCAE v. 3.0)
* History of clinically relevant psychiatric disability, precluding informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Actual)
Dates: Start 2010-10; Primary Completion 2017-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Relapse Free Survival | 3-years

SECONDARY OUTCOMES:
Overall Survival | 3-years
Safety Profil according to NCI-CTAE v 3.0 | q2w
  Percentage (%) of treatments delays and interaptions in each arm Percentage (%) of dose received versus planned dose in each arm

CONTACTS AND LOCATIONS:
Overall Officials: John Souglakos, MD, Principal Investigator — University Hospital of Crete, Dep of Medical Oncology; Vassilis Georgoulias, MD, Study Chair — University Hospital of Crete, Dep of Medical Oncology
Locations (1):
- University Hospital of Crete, Dep of Medical Oncology, Heraklion, Greece

REFERENCES:
- [Derived] Gallois C, Shi Q, Meyers JP, Iveson T, Alberts SR, de Gramont A, Sobrero AF, Haller DG, Oki E, Shields AF, Goldberg RM, Kerr R, Lonardi S, Yothers G, Kelly C, Boukovinas I, Labianca R, Sinicrope FA, Souglakos I, Yoshino T, Meyerhardt JA, Andre T, Papamichael D, Taieb J. Prognostic Impact of Early Treatment and Oxaliplatin Discontinuation in Patients With Stage III Colon Cancer: An ACCENT/IDEA Pooled Analysis of 11 Adjuvant Trials. J Clin Oncol. 2023 Feb 1;41(4):803-815. doi: 10.1200/JCO.21.02726. Epub 2022 Oct 28. PMID 36306483
- [Derived] Iveson TJ, Sobrero AF, Yoshino T, Souglakos I, Ou FS, Meyers JP, Shi Q, Grothey A, Saunders MP, Labianca R, Yamanaka T, Boukovinas I, Hollander NH, Galli F, Yamazaki K, Georgoulias V, Kerr R, Oki E, Lonardi S, Harkin A, Rosati G, Paul J. Duration of Adjuvant Doublet Chemotherapy (3 or 6 months) in Patients With High-Risk Stage II Colorectal Cancer. J Clin Oncol. 2021 Feb 20;39(6):631-641. doi: 10.1200/JCO.20.01330. Epub 2021 Jan 13. PMID 33439695
- [Derived] Souglakos J, Boukovinas I, Kakolyris S, Xynogalos S, Ziras N, Athanasiadis A, Androulakis N, Christopoulou A, Vaslamatzis M, Ardavanis A, Emmanouilides C, Bompolaki I, Kourousis C, Makrantonakis P, Christofyllakis C, Athanasiadis E, Kentepozidis N, Karampeazis A, Katopodi U, Anagnosopoulos A, Papadopoulos G, Prinarakis E, Kalisperi A, Mavroudis D, Georgoulias V. Three- versus six-month adjuvant FOLFOX or CAPOX for high-risk stage II and stage III colon cancer patients: the efficacy results of Hellenic Oncology Research Group (HORG) participation to the International Duration Evaluation of Adjuvant Chemotherapy (IDEA) project. Ann Oncol. 2019 Aug 1;30(8):1304-1310. doi: 10.1093/annonc/mdz193. PMID 31228203